CLINICAL TRIAL: NCT05522153
Title: A Single Blinded Randomized Control Trial Comparing the Use of ARISTA Polysaccharide Hemostat in Total Knee Arthroplasty (TKA)
Brief Title: Arista Hemostatic Powder for Total Knee Post Operative Outcomes Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virtua Health, Inc. (Other)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: virtuamcmillan1
Record Dates: First submitted 2022-04-25; First posted 2022-08-30 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Arista

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant
Masking Description: patients are blinded as to their randomization group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arista group (Experimental): this group of randomized patients will receive 5 grams of arista hemostatic powder intra-operatively in their wound in addition to 1 gram of IV transexemic acid prior to incision
  Interventions: Drug: Arista
- control group (No Intervention): this group of randomized patients will receive just the 1 gram of IV transexemic acid prior to incision

INTERVENTIONS:
Drug: Arista — hemostatic powder
  Arms: Arista group

SUMMARY:
To examine in Arista hemostatic powder results in less post-total knee arthroplasty blood loss, hematoma formation, and improved range of motion when compared to patients who did not receive the product.

DETAILED DESCRIPTION:
Patients will be recruited from the Hospital for Special Surgery and Our Lady of Lourdes Programs. Patients will be prospectively enrolled when Institutional Review Board (IRB) approval is obtained. All patients will be undergoing a primary unilateral total knee arthroplasty for a diagnosis of osteoarthritis. Once enrolled in the study, each patient will be randomized into one of two groups. Group A will undergo a TKA utilizing Arista MPH ® intra-operatively. Group B will undergo a TKA without Arista MPH ®. All patients will receive a baseline IV dose of tranexamic acid per weight based guidelines prior to incision.

A thigh tourniquet will be utilized from prior to incision until wound closure is complete. Arista MPH ® will be used intra-operatively. A 5 gram vial of Arista MPH will be the standard of use. ARISTA will be used in accordance with the instructions for use. Additional need for Arista MPH ® usage during the case will be permitted and recorded. Standard electrocautory will be permitted, however additional thermal devices intended for hemostatic control will not be utilized.

Pre-operative hemoglobin, hematocrit, PT, PTT, and INR will be per standard institutional protocol within 30 days of surgery. The hemoglobin and hematocrit will be repeated 24 hours after the procedure per standard physician protocol. IV fluids administered pre-op, intra-op and post op for the first 24 hours will be recorded. Administration of any blood products from the time of incision until 90 days post-op will be recorded. Blood loss will be calculated via standard HSS. Drains will not be utilized.

The transfusion criteria is: a hemoglobin level of <8 g/dL or a hemoglobin level of <10 g/dL in a patient with symptomatic anemia or deemed at high risk because of notable underlying cardiac comorbidities. Blood will be administered 1 unit at a time, and the presence of symptoms or signs was reassessed.

Pre-operative thigh circumference will be measured on the day of the surgery. For standardization, the circumference will be recorded 15 cm proximal to the superior pole of the patella. Post-operatively the thigh circumference will be measured at 24 hours, post-operative day 14 +/- 4 days, and post operatively at 3 months +/- 1 week.

Post-operative knee range of motion will be recorded at 24 hours, post-operative day 14 +/- 4 days, and post-operatively at 3 months +/- 1 week.

Pre-operative and post-operative day 14 (+/- 4 days) and post-operative 3 months (+/- 1 week) knee society short form scores will be collected All post-operative adverse events related to the procedure will be recorded. These invents include, but are not limited to: readmission, infection, prosthesis loosening, wound dehiscence, and wound drainage.

All data will be de-identified and securely maintained in an IRB approved manner.

ELIGIBILITY:
Inclusion Criteria:

* • They willingly desire to participate and signed the informed consent

  * Are between the ages of 18 and 100 years of age
  * Have the mental capacity to provide consent
  * Are undergoing a primary unilateral total knee arthroplasty

Exclusion Criteria:

* • allergy to Arista MPH®

  * allergy to tranexamic acid
  * preoperative hepatic or renal dysfunction
  * serious cardiac or respiratory disease including coronary artery stent placement
  * congenital or acquired coagulopathy as evidence by INR > 1.4 or PTT > 1.4 times normal
  * thrombocytopenia as identified by a preoperative platelet count of < 150,000/mm3
  * history of thromboembolic disease
  * pregnant or breast feeding
  * donated preoperative autologous blood
  * diagnosis of inflammatory arthritis
  * a preoperative hemoglobin < 10 g/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Virtua Health System, Marlton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arista Group | Control Group
Started | 31 | 30
Completed | 31 | 28
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arista Group | Control Group | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (8.0) | 65.9 (8.4) | 66.31 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 14 | 10 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 25 | 20 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Blood Loss
Description: Calculated on standard hospital protocol
Time Frame: Time of incision until 90 days post-op
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | Arista Group | Control Group
Number analyzed (Participants) | 31 | 30
cubic centimeters | 122.6 (25.3) | 133.3 (42.2)

2. Secondary Outcome: Thigh Circumference
Description: Thigh circumference measurement 15 cm above the top of the patella
Time Frame: 3 months post op
Population: 61 patients were consented however some did not continue to the 3 month post op timepoint and therefore their data was not collected or analyzed.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Arista Group | Control Group
Number analyzed (Participants) | 30 | 26
centimeters | 50.6 (6.7) | 54 (6.9)

3. Secondary Outcome: Range of Motion
Description: Measured in degrees
Time Frame: 3 months post op
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Arista Group | Control Group
Number analyzed (Participants) | 30 | 24
Degrees | 117.8 (9.6) | 114.3 (11.7)

ADVERSE EVENTS:
Time Frame: Enrollment to 90 Days post-op
Arm/Group | Arista Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/31 | 2/28
Other Adverse Events (participants affected / at risk) | 2/31 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arista Group (N=31) | Control Group (N=28)
Readmission due to pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) — Readmission due to pain, unrelated to study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arista Group (N=31) | Control Group (N=28)
Infection (Infections and infestations) | 2 (2) | 0 (0) — Infection post procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT05522153/Prot_000.pdf
  • Informed Consent Form (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT05522153/ICF_001.pdf